CLINICAL TRIAL: NCT01582425
Title: A Phase 1, Open-Label, Sequential Study of the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Methadone in Healthy Adult Subjects
Brief Title: Drug Interaction Study of Isavuconazole and Methadone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0027
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Methadone; Healthy Volunteers
Keywords: isavuconazole; methadone; Healthy Volunteers; BAL8557
MeSH Terms: interventions — isavuconazole; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and methadone (Experimental): Single dose of methadone on Days 1 and 20, isavuconazole 3 times a day (TID) on Days 16-17 as a loading dose, isavuconazole once a day (QD) on Days 18-28
  Interventions: Drug: Isavuconazole; Drug: Methadone

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557; BAL4815
Drug: Methadone — oral
  Other Names: Dolopine

SUMMARY:
The primary purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics (PK) of methadone after single dose administration. The secondary purpose is to assess the safety and tolerability of isavuconazole alone and in combination with methadone.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be ≤ upper limit of normal and total bilirubin must be ≤ 1.5 mg/dL
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a positive result for hepatitis C antibodies, hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products including methadone or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics (PK) of plasma for R-methadone and S-methadone: AUClast, AUCinf, and Cmax | Days 1 and 20
  Area under the curve (AUC) from time of dosing to last quantifiable concentration (AUClast ), AUC from time 0 extrapolated to infinity (AUCinf), maximum concentration (Cmax)

SECONDARY OUTCOMES:
Composite of pharmacokinetics (PK) of plasma for R-methadone and S-methadone : tmax,t1/2, Vz/F, and CL/F | Days 1 and 20
  Time to attain Cmax (tmax) , apparent terminal elimination half-life (t1/2), apparent volume of distribution (Vz /F), and apparent body clearance after oral dosing (CL/F)
PK of plasma isavuconazole: trough concentration (Ctrough) | Days 18 and Days 21 through 29
Composite of PK of plasma isavuconazole: AUC during the time interval between consecutive dosing (AUCtau), Cmax, and tmax | Days 19 and 20
Safety assessed by recording of adverse events, laboratory evaluations, electrocardiograms (ECGs) and vital signs | Up to Day 36

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, LLC, Glendale, California, United States